CLINICAL TRIAL: NCT06708520
Title: A Study to Investigate Pharmacokinetics and Safety of Rupatadine (10 mg) and Its Active Metabolites in Participants With Renal Impairment Compared to Matched Control Participants With Normal Renal Function
Brief Title: Pharmacokinetics and Safety of Rupatadine in Participants With Renal Impairment Compared to Control Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Noucor Health S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DC09RUP/1/21
Record Dates: First submitted 2022-04-27; First posted 2024-11-27 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — rupatadine

STUDY DESIGN:
Intervention Model Description: Phase 1, single dose, open-label, parallel group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Renal impairement mild (Experimental)
  Interventions: Drug: Rupatadine
- Renal impairement moderate (Experimental)
  Interventions: Drug: Rupatadine
- Renal impairement severe (Experimental)
  Interventions: Drug: Rupatadine
- Renal normal functions (Experimental)
  Interventions: Drug: Rupatadine

INTERVENTIONS:
Drug: Rupatadine — 10 mg tablets
  Other Names: Pafinur

SUMMARY:
The purpose of this study is to assess the PK, tolerability, and safety of rupatadine (10 mg) and its active metabolites in participants with renal impairment compared to matched control participants with normal renal function.

The study duration will be up to 40 days, including Screening, Baseline, Study Period, and EOS visit assessments.

Rupatadine 10 mg tablet will be administered as single dose.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, parallel group study comparing the PK after administration of a single 10 mg dose of rupatadine to participants with renal impairment with matched control participants with normal renal function (matched in terms of gender, age, and body weight).

For each participant, the study visits will consist of a Screening Period (Day -28 to Day -2), a Baseline evaluation (Day -1), a single dose treatment period (Day 1) and an End of Study (EOS) Visit (Day 12 for subjects with renal impairment and Day 8 for subjects with normal real function). Additionally, from Day 2 to EOS participants will go back to the clinic for blood drawing according to schedule.

Participants who meet the eligibility criteria at Screening and Baseline will be enrolled into the study.

All Baseline safety evaluation results must be reviewed prior to dosing. Participants will be domiciled at the clinic from Day -1 until 24 hours after dosing on Day 1 (Day 2).

On Day 1, participants will receive a single dose of rupatadine 10 mg after an overnight fast of 10 hours and will continue to fast for 4 hours post-dose.

Participants with renal impairment will undergo sequential PK sampling over the following 264 hours along with other safety assessments. Participants with normal renal function will undergo sequential PK sampling over the following 144 hours along with other safety assessments.

The participant groups will be consecutively enrolled into the study. Enrollment of participants with mild, moderate, and severe renal impairment will be staggered, so that dosing of participants with mild renal impairment will be started first. Dosing of the next group will be started only after evaluation of blood PK, safety and tolerability data until 72 hours post dose of at least six participants with renal impairment from the previous group and after the assessment of safety and tolerability results are judged to be satisfactory by the Safety Committee.

An EOS assessment will occur 7 days after the administration of rupatadine in the participants with normal renal function and 11 days after in renal impaired participants.

The total study duration, including Screening, Baseline, Study Period, and EOS assessments, is up to approximately 40 days.

ELIGIBILITY:
Inclusion Criteria:

Participants with normal renal function and participants with mild, moderate, or severe renal impairment who meet the following criteria will be considered eligible to participate in the clinical study:

1. Participant understands the study procedures and agrees to participate in the study by giving written informed consent prior to any study-mandated procedure.
2. Able to communicate well with the Investigator, to understand and comply with the study requirements.
3. Willing to comply with study restrictions stated in Section 5.3 (lifestyle considerations).
4. Male or female Caucasian subjects, between 18 and 75 years (inclusive) of age.
5. Body mass index (BMI) is between 18 to 35 kg/m2 at Screening.
6. Women of childbearing potential (WoCBP) must have a negative serum pregnancy test at Screening, a negative urine pregnancy test on Day -1, and agree to consistently and correctly use (from 30 days prior to dosing, during the entire study, and for at least 30 days after dosing), a highly effective method of contraception (i.e., failure rate of < 1%) (Section 10.4 [Appendix 4]). Such methods include:

   - Hormonal contraceptives: combined (estrogen- and progesterone-containing) contraception associated with inhibition of ovulation using oral, intravaginal, or transdermal route of administration.

   Note: If a hormonal contraceptive is used, it must be initiated at least 30 days before dosing.
   * Intrauterine device.
   * Intrauterine hormone-releasing system.
   * Bilateral tubal occlusion.
   * Vasectomized partner, provided that the partner is the sole sexual partner and that the vasectomized partner has received medical assessment of the surgical success.
   * Sexual abstinence, defined as refraining from heterosexual intercourse from 30 days prior to dosing up to at least 30 days after dosing, if this is the preferred and usual lifestyle of the subject.

   WoCBP must also agree not to donate ova from the time of informed consent until 30 days after dosing
7. Women of non-childbearing potential (WoNCBP), i.e., postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by a follicular stimulating hormone [FSH] test), with previous bilateral salpingectomy, bilateral salpingo-oophorectomy or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, uterine agenesis (Section 10.4 [Appendix 4]).
8. Male participants are infertile, vasectomized (who has received medical assessment of the surgical success) or must agree to abstain from, or to use a condom, during heterosexual intercourse with a woman of childbearing potential (Section 10.4 [Appendix 4]).
9. Male participants must agree not to donate sperm, from the time of informed consent until 30 days after dosing.
10. Negative test results for anti-Human Immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), Hepatitis B surface antigen (HBsAg) and anti-Hepatitis Cvirus antibodies (anti-HCVAb).
11. Participant agrees to refrain from consuming grapefruit juice, grapefruits, and grapefruitcontaining products from at least 7 days before the dose administration, and until the EOS Visit.
12. Able to tolerate venipuncture

    For participants with mild, moderate, or severe renal impairment, the following criteria must be met in addition:
13. Participants with impaired renal function should be hemodynamically stable.
14. Diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in renal function) renal impairment.
15. Estimated GFR must range from:

    1. 15-29 mL/min (severe renal impairment) or
    2. 30-59 mL/min (moderate renal impairment) or
    3. 60-89 mL/min (mild renal impairment) determined by the Cockcroft-Gault equation, at the Screening Visit.
16. Stable concomitant medications for at least 21 days prior to dosing and up to the EOS visit.
17. Systolic blood pressure (SBP) 100-180 mmHg, diastolic blood pressure (DBP) 50-105 mmHg and pulse rate 60-100 bpm (inclusive), measured on the same arm, after 5 min in the supine position at Screening and Baseline.

    For participants with normal renal function, the following criteria must be met in addition:
18. No clinically relevant diseases captured in medical history at Screening.
19. No clinically relevant abnormalities on physical examination at Screening and Baseline.
20. No clinically relevant abnormalities on clinical laboratory tests at Screening.
21. Normal renal function confirmed by estimated creatinine clearance (eCLcr) ≥ 90 mL/min, as determined by the Cockcroft-Gault equation, at Screening.
22. Weight within ±15% to his/her matched participant(s) enrolled in the study.
23. Biological sex matched to his/her matched participant(s) enrolled in the study.
24. Age within ±10 years to his/her matched participant(s) enrolled in the study.
25. Normal BP measured on the same arm, after 5 min in the supine position at Screening and Baseline defined as:

    * SBP 90-140 mmHg, DBP 60-90 mmHg, and pulse rate 60-100 bpm (inclusive) for subjects < 65 years of age.
    * SBP 95-160 mmHg, DBP 65-95 mmHg, and pulse rate 60-100 bpm (inclusive) for subjects ≥ 65 years of age.

Exclusion Criteria:

Participants with normal renal function and participants with mild, moderate, or severe renal impairment who meet one or more of the following criteria will not be considered eligible to participate in the clinical study:

1. Pregnant or lactating women.
2. Participant is unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for the EOS Visit and improbability of completing the clinical study.
3. Any psychological, emotional problems, any disorders or resultant therapy that is likely to invalidate informed consent, or limit the ability of the participant to comply with the protocol requirements
4. History of hypersensitivity to rupatadine, desloratadine or any of the excipients, or to medicinal products with similar chemical structures.
5. History of clinically significant lactose, galactose, or fructose intolerance.
6. Any clinically relevant acute or chronic disease which could jeopardize the safety of the participant or impact the validity of the study results.
7. Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
8. Participation in another clinical trial with an experimental drug within 2 months or 5 halflives (whichever is longer) before the Screening or in more than 2 clinical studies within 1 year prior to Screening.
9. History or presence of clinically significant angioedema.
10. Use of caffeine-containing beverages exceeding 800 mg per day (Section 5.3.2) at Screening.
11. Nicotine consumption (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) from 48 h prior to Baseline (Day -1) until discharge from confinement (Day 2).
12. Positive test result for urine alcohol and drugs of abuse (amphetamines, benzodiazepines, cannabinoids, cocaine and opiates) at Screening and Baseline.

    Note: Subjects receiving stable treatment of methadone and benzodiazepines will be allowed to be enrolled in the study even if the urine drug screen test is positive.
13. History of heart, kidney or liver transplantation.
14. History of stroke, chronic seizures, or major neurological disorder.
15. Active malignant neoplastic disease or carcinoma (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment.
16. Intake of any creatine supplement from Screening to EOS.
17. Use of any of the following 2 weeks prior to investigational medicinal product (IMP) administration or 5 half-lives, whichever is longer:

    1. Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism (e.g., azole antifungals [ketoconazole, itraconazole, fluconazole, Posaconazole, voriconazole], macrolide antibiotics [erythromycin, clarithromycin], diltiazem, human immunodeficiency virus (HIV) protease inhibitors, nefazodone, rifampicin, phenytoin, dexamethasone, troglitazone, and barbiturates)
    2. CYP3A4 substrates with a narrow therapeutic index (e.g. ciclosporin, tacrolimus, sirolimus, everolimus, cisapride)
    3. Desloratadine
18. Clinically significant abnormalities on ECG repolarization (QTcF > 450 ms in males and >470 ms in females) at Screening.
19. Loss of 250 mL or more blood within 3 months prior to screening.

    For participants with mild, moderate or severe renal impairment the additional criteria must not be met:
20. Fluctuating or rapidly deteriorating renal function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of renal impairment within the Screening Period.
21. Participants requiring dialysis.
22. History or clinical evidence of any disease (except for renal impairment) and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of rupatadine, and/or the ability to complete the study.

    For participants with normal renal function, the additional criteria must not be met:
23. History or presence of a clinically relevant abnormality in any organ system, that is incapacitating, requires hospitalization, or in the opinion of the investigator makes the participant ineligible for enrollment in the study.
24. History or clinical evidence of any disease and/or existence of any surgical or medical condition that might have interfered with the absorption, distribution, metabolism, or excretion of rupatadine (appendectomy and herniotomy are allowed, cholecystectomy is not allowed).
25. Intake of any prescribed medication (including vaccines) including over-the-counter (OTC) medication (including herbal and dietary supplements such as St John's Wort, homeopathic preparations, vitamins and minerals) that could affect the outcome of the study as judged by the Investigator, within 14 days before the administration of the IMP or less than 5 times the half-life of that medication, whichever is longer (excluding contraceptives and hormone replacement therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to last timepoint (AUC0-t) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to last timepoint (AUC0-t), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to infinity (AUC0-inf), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Peak plasma concentration (Cmax) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the peak plasma concentration (Cmax), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Time of maximum plasma concentration (tmax) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the time of maximum plasma concentration (tmax) of rupatadine, of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Plasma fraction unbound (fu) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the plasma fraction unbound (fu), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Terminal elimination rate constant (kel) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the terminal elimination rate constant (kel), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Terminal half-life (t1/2) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the terminal half-life (t1/2), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Apparent total plasma clearance (CL/F) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the apparent total plasma clearance (CL/F), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Apparent volume of distribution during terminal phase (Vz/F) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the apparent volume of distribution during terminal phase (Vz/F), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Apparent non-renal clearance (CLNR/F) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the apparent non-renal clearance (CLNR/F), calculated as apparent total clearance - renal clearance, of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Renal clearance (CLR) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the renal clearance (CLR), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Amount excreted unchanged (Ae) in urine of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the amount excreted unchanged (Ae) in urine, of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Fraction excreted in urine (fe; fe%) of rupatadine | 12 days
  To assess the pharmacokinetics (PK), including the fraction excreted in urine (fe; fe%), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Peak plasma concentration (Cmax) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the peak plasma concentration (Cmax) , of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Area under the plasma concentration-time curve from time zero to last timepoint (AUC0-t) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to last timepoint (AUC0-t), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to infinity (AUC0-inf), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Time of maximum plasma concentration (tmax) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the time of maximum plasma concentration (tmax) , of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Terminal half-life (t1/2) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the terminal half-life (t1/2), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Renal clearance (CLR) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the renal clearance (CLR), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)
Metabolic ratio (MR) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 12 days
  To assess the pharmacokinetics (PK), including the metabolic ratio (MR), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to last timepoint (AUC0-t) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the area under the plasma concentration-time curve from time zero to last timepoint (AUC0-t)
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the area under the plasma concentration-time curve from time zero to infinity (AUC0-inf)
Peak plasma concentration (Cmax) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the peak plasma concentration (Cmax)
Time of maximum plasma concentration (tmax) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the time of maximum plasma concentration (tmax)
Terminal elimination rate constant (kel) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the terminal elimination rate constant (kel)
Terminal half-life (t1/2) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the terminal half-life (t1/2)
Apparent total plasma clearance (CL/F) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the apparent total plasma clearance (CL/F)
Renal clearance (CLR) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the renal clearance (CLR)
Apparent non-renal clearance (CLNR/F) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the apparent non-renal clearance (CLNR/F)
Apparent Volume of Distribution During Terminal Phase (V/F) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the apparent Volume of Distribution During Terminal Phase (V/F)
Incidence of treatment-emergent adverse events (TEAEs) | 12 days
  To determine the safety and tolerability, including the incidence of treatment-emergent adverse events (TEAEs), of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants with normal renal function (control).
Change from Baseline in electrocardiogram (ECG) parameters | 12 days
  To determine the safety and tolerability, including the change from Baseline in electrocardiogram (ECG) parameters, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants
Change from Baseline in vital signs | 12 days
  To determine the safety and tolerability, including the change from Baseline in vital signs, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants
Change from Baseline in selected safety laboratory parameters | 12 days
  To determine the safety and tolerability, including the change from Baseline in selected safety laboratory parameters, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants
Change from Baseline in body weight | 12 days
  To determine the safety and tolerability, including the change from Baseline in body weight, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe renal impairment in comparison to participants

OTHER OUTCOMES:
The relationship between renal function (estimated glomerular filtration rate [eGFR] using modification of diet in renal disease equation) and PK parameters (AUC0-t and Cmax) for rupatadine and its metabolites in terms of plasma concentrations | 12 days
  The relationship between renal function (estimated glomerular filtration rate [eGFR] using modification of diet in renal disease equation) and PK parameters (AUC0-t and Cmax) for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Guimarães, Principal Investigator — Blueclinical Investigacao E Desenvolvimento Em Saude Lda.; Rosa Maria Príncipe, MD, Principal Investigator — Hospital Pedro Hispano; Daniela Machado Lopes, MD, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia/Espinho; Dolores Ochoa Mazarro, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Ana Maria Aldea Perona, MD, Principal Investigator — Municipal Institute Of Medical Investigation; Jordi Soler Majoral, MD, Principal Investigator — Germans Trias i Pujol Hospital; Rosa Maria Antonijoan Arbós, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (7):
- Portugal (3):
  - Centro Hospitalar De Vila Nova De Gaia Espinho, Gaia
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Blueclinical Investigacao E Desenvolvimento Em Saude Lda., Porto
- Spain (4):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Municipal Institute Of Medical Investigation, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario De La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billah MM, Chapman RW, Egan RW, Gilchrest H, Piwinski JJ, Sherwood J, Siegel MI, West RE Jr, Kreutner W. Sch 37370: a potent, orally active, dual antagonist of platelet-activating factor and histamine. J Pharmacol Exp Ther. 1990 Mar;252(3):1090-6. PMID 2319461
- [Background] Eiser NM, Mills J, Snashall PD, Guz A. The role of histamine receptors in asthma. Clin Sci (Lond). 1981 Apr;60(4):363-70. doi: 10.1042/cs0600363. PMID 7249528
- [Background] Cuss FM, Dixon CM, Barnes PJ. Effects of inhaled platelet activating factor on pulmonary function and bronchial responsiveness in man. Lancet. 1986 Jul 26;2(8500):189-92. doi: 10.1016/s0140-6736(86)92489-x. PMID 2873440
- [Background] Henocq E, Vargaftig BB. Accumulation of eosinophils in response to intracutaneous PAF-acether and allergens in man. Lancet. 1986 Jun 14;1(8494):1378-9. doi: 10.1016/s0140-6736(86)91683-1. No abstract available. PMID 2872485
- [Background] Piwinski JJ, Wong JK, Green MJ, Ganguly AK, Billah MM, West RE Jr, Kreutner W. Dual antagonists of platelet activating factor and histamine. Identification of structural requirements for dual activity of N-Acyl-4-(5,6-dihydro-11H-benzo [5,6]cyclohepta-[1,2-b]pyridin-11-ylidene)piperidines. J Med Chem. 1991 Jan;34(1):457-61. doi: 10.1021/jm00105a069. No abstract available. PMID 1671420
- [Background] Prescott SM, Zimmerman GA, McIntyre TM. The production of platelet-activating factor by cultured human endothelial cells: Regulation and function. In Platelet-activating factor and related lipid mediators. Snyder F, Ed. New York: Plenum Press, 1987: 323-340.
- [Background] Katiyar S, Prakash S. Pharmacological profile, efficacy and safety of rupatadine in allergic rhinitis. Prim Care Respir J. 2009 Jun;18(2):57-68. doi: 10.3132/pcrj.2008.00043. PMID 18695846
- [Background] Mullol J, Bousquet J, Bachert C, Canonica WG, Gimenez-Arnau A, Kowalski ML, Marti-Guadano E, Maurer M, Picado C, Scadding G, Van Cauwenberge P. Rupatadine in allergic rhinitis and chronic urticaria. Allergy. 2008 Apr;63 Suppl 87:5-28. doi: 10.1111/j.1398-9995.2008.01640.x. PMID 18339040
- [Background] Queralt M, Brazis P, Merlos M, de Mora F, Puigdemont A. In vitro inhibitory effect of rupatadine on histamine and TNF-alpha release from dispersed canine skin mast cells and the human mast cell line HMC-1. Inflamm Res. 2000 Jul;49(7):355-60. doi: 10.1007/PL00000216. PMID 10959557
- [Background] Merlos M, Ramis I, Balsa D, Queralt M, Brazís P, Puigdemont A. Inhibitory effect of rupatadine on TNF-a release from human monocytes and mast cell lineHMC-1. J.Allergy Clin. Immunol. 2000 105(Suppl.1): S62.
- [Background] Bartra J, Valero AL, del Cuvillo A, Davila I, Jauregui I, Montoro J, Mullol J, Sastre J. Interactions of the H1 antihistamines. J Investig Allergol Clin Immunol. 2006;16 Suppl 1:29-36. No abstract available. PMID 17357375
- [Background] del Cuvillo A, Mullol J, Bartra J, Davila I, Jauregui I, Montoro J, Sastre J, Valero AL. Comparative pharmacology of the H1 antihistamines. J Investig Allergol Clin Immunol. 2006;16 Suppl 1:3-12. No abstract available. PMID 17357372
- [Background] Olkkola KT, Ahonen J. Midazolam and other benzodiazepines. Handb Exp Pharmacol. 2008;(182):335-60. doi: 10.1007/978-3-540-74806-9_16. PMID 18175099
- [Background] Picado C. Rupatadine: pharmacological profile and its use in the treatment of allergic disorders. Expert Opin Pharmacother. 2006 Oct;7(14):1989-2001. doi: 10.1517/14656566.7.14.1989. PMID 17020424
- [Background] Izquierdo I, Merlos M, Garcia-Rafanell J. Rupatadine: a new selective histamine H1 receptor and platelet-activating factor (PAF) antagonist. A review of pharmacological profile and clinical management of allergic rhinitis. Drugs Today (Barc). 2003 Jun;39(6):451-68. doi: 10.1358/dot.2003.39.6.799450. PMID 12944997
- [Background] Keam SJ, Plosker GL. Rupatadine: a review of its use in the management of allergic disorders. Drugs. 2007;67(3):457-74. doi: 10.2165/00003495-200767030-00008. PMID 17335300
- [Background] European Medicines Agency. Committee for Medicinal Products for Human Use Guidance: Guideline on the Investigation of Drug Interactions. 21 June 2012.
- [Background] Rupatadine Investigator's Brochure, dated 21 Sep 2021.
- [Background] Food and Drug Administration Guidance: Pharmacokinetics in Patients with Impaired Renal Function: Study Design, Data Analysis, and Impact on Dosing . September 2020.
- [Background] European Medicines Agency. Committee for Medicinal Products for Human Use Guidance: Guideline on the evaluation of the pharmacokinetics of medicinal products in patients with decreased renal function. December 2015.
- [Background] FDA Guidance: Conduct of Clinical Trials of Medical Products During the COVID-19 Public Health Emergency-Guidance for Industry, Investigators, and Institutional Review Boards: August 2021.
- [Background] DMID ALCOAC Checklist V2.0 29 January 2020.
- See also: Summary of Product Characteristics (SmPC) for rupatadine — https://www.medicines.org.uk/emc/product/2501/smpc#gref